CLINICAL TRIAL: NCT05466071
Title: Safety and Efficacy of Tenofovir Alafenamide to Prevent Mother-to-child Transmission of Hepatitis B Virus in Middle/Late Pregnancies With High Hepatitis B Virus DNA Load: A Prospective Multicenter Cohort Study
Brief Title: Safety and Efficacy of TAF to Prevent MTCT of HBV in Middle/Late Pregnancies With High HBV DNA Load
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xingfei Pan (Other)
Responsible Party: Sponsor-Investigator, Xingfei Pan, Director of Department of Infectious Diseases, The Third Affiliated Hospital of Guangzhou Medical University
Organization: The Third Affiliated Hospital of Guangzhou Medical University (Other)
Other Study IDs: LCYJ-2021-005
Record Dates: First submitted 2022-07-07; First posted 2022-07-20 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Chronic Hepatitis b; Pregnancy Related
Keywords: Tenofovir Alafenamide; Safety and Efficacy; Mother-to-Child Transmission; High HBV DNA Load
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TAF group: Patients who take TAF during pregnancy.
- TDF group: Patients who take TDF during pregnancy.

SUMMARY:
Mother-to-child transmission (MTCT) is still the main transmission route of HBV in high-endemic areas, such as China, sub-Saharan Africa, etc. Some infants born of mothers with high HBV DNA load (≥2×10^5 IU/ml) are still infected with HBV even if these infants receive the combined immunization on time. Therefore, guidelines including AASLD and EASL recommend that pregnant women with high HBV DNA load should take antiviral drugs (tenofovir disoproxil fumarate or telbivudine) to reduce MTCT of HBV from gestation 24-28 weeks.

However, side effects of TDF on infants are reported. For example, neutropenia and the decrease of bone mineral density are found in early age infants who are ever exposed to TDF during their fetal life.

Tenofovir alafenamide (TAF), a new prodrug of tenofovir (TFV), has a higher antiviral potency, a higher peripheral blood mononuclear cell (PBMC) intracellular tenofovir diphosphate (TFV pp) level and a lower plasma TFV concentration. As the successor of TDF, the dose of TAF that is took orally every day is approximately 1/10 of TDF. TAF has a much lower risk of kidney toxicity and has almost no effect on the bone mineral density. TAF has been approved and recommended as the first-line drug to treat patients with chronic hepatitis B (CHB) by AASLD, EASL, etc. However, there are relatively few data of TAF on pregnancies with high HBV DNA load. It is urgently to clarify the safety and efficacy of TAF on interrupting MTCT of HBV in pregnancies with high HBV DNA load.

In the present study, the investigators enroll middle/late pregnancies with high HBV DNA load(≥2×10^5 IU/ml). The participants are randomly divided into two groups. Then the participants are treated with TAF or TDF respectively. All enrolled participants are followed-up for 2 years. Objectives of the present study are as follows:

A. To clarify safety and efficacy of TAF on interrupting MTCT of HBV in middle/late pregnancies with high HBV DNA load.

B. To clarify effects of TAF on obstetric complications in middle/late pregnancies with CHB.

C. To clarify effects of TAF on birth defects of infants born in mothers with CHB.

D. To clarify the change of virology and biochemistry indexes in women with CHB during pregnancy and postpartum.

E. To clarify effects of TAF treatment on participants. F. To clarify growth parameters of the infants exposed to TAF during their fetal life.

G. To clarify the pharmacokinetics of TAF in pregnant populations.

ELIGIBILITY:
Inclusion Criteria:

* Age of 20-40 years.
* Positive for HBsAg ≥6 months.
* HBV DNA load of ≥ 2×10^5 IU/ml.
* Gestation 24-28 weeks .
* Pregnancies are orally administrated with TAF (25mg/day) or TDF (300mg/day) from 24-28 weeks of gestation.
* The good compliance of patients.

Exclusion Criteria:

* Patients with antibodies against HIV, HCV, HDV, or other forms of chronic liver disease.
* Evidence of hepatocellular carcinoma, decompensated liver disease, auto-immune hepatitis, or significant renal, cardiovascular, respiratory or neurological comorbidity.
* Concurrent treatment with nephrotoxic drugs, glucocorticoids, cytotoxic drugs, nonsteroidal anti-inflammatory drugs, or immune modulators.
* Ultra-sonographic evidence of fetal deformity, abnormal fetal development or placental abnormality.
* Clinical signs of threatened miscarriage.
* History of complication of pregnancy.
* History of nucleoside analogues (NA) treatment.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: We enroll Child-bearing age women with chronic HBV infection, who already become middle/late pregnancy, and visit in 3 hospitals (The Third Affiliated Hospital of Guangzhou Medical University, People's Hospital of Guangzhou Huadu District and He Xian Memorial Hospital of Guangzhou Panyu District).
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of interrupting MTCT | During 7-12 months after birth
  The proportion of HBV infection in the infants at 1 year of age.
  Testing for HBsAg in the infants between 7 and 12 months of age.
HBV DNA load in pregnancies | After enrollment and up to delivery
  HBV DNA load is measured during 24-28 weeks of gestation and at birth, respectively.
ALT levels in pregnancies | After enrollment and up to delivery
  ALT levels are measured every month during pregnancy.
HBeAg conversion rate in pregnancies | After enrollment and up to delivery
  HBeAg is measured every 6 months during pregnancy.

SECONDARY OUTCOMES:
Mode of delivery. | At the time of delivery
  Recording the mode of delivery (vaginal delivery or cesarean delivery), and what kind of anesthesia (general anesthesia or combined spinal/epidural anesthesia) is used in the cesarean delivery.
The proportion of birth defects in the infants at 1 month age. | Up to 1 month after birth
  Measuring which kinds of congenital abnormality the infants have.
Head circumferences of infants | Once a year up to 3 years old after birth
  Head circumferences of infants are measured and analyzed.
Weights of infants | Once a year up to 3 years after birth
  Weights of infants are measured and analyzed.
Heights of the infants | Once a year up to 3 years after birth
  Heights of the infants are measured and analyzed.
Denver Developmental Screening Test of infants | Once a year up to 3 years after birth
  Denver Developmental Screening Test of infants is measured and analyzed.
HBV DNA load in postpartum mothers | Up to 2 years after delivery
  HBV DNA load is measured every 6 months postpartum.
ALT levels in postpartum mothers | Up to 2 years after delivery
  ALT levels are measured every month during the first 3 months postpartum and every 6 months from the fourth month postpartum.
HBeAg conversion rate in postpartum mothers | Up to 2 years after delivery
  HBeAg is measured every 6 months after delivery.
Liver function of women with CHB | Up to 2 years after delivery
  Liver function is measured every 6 months postpartum.
Liver ultrasound test of women with CHB | Up to 2 years after delivery
  Liver ultrasound is performed every 6 months postpartum.
The blood drug concentration of TAF in pregnancies | Day 5 up to day 40 after the administration of TAF
  After the administration of TAF to pregnant women, 4 ml of upper extremity venous drug-containing blood is collected between 30 and 60 minutes before the next taking TAF at the 5th, 12th, 19th, 26th, 33rd, and 40th days, respectively. After a series of laboratory processes, the supernatant is taken for HPLC-MS/MS analysis, and the blood drug concentration at each time point is calculated according to the standard curve.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Affiliated Hospital, Guangzhou Medical University, Guangzhou, Guangdong, China